CLINICAL TRIAL: NCT02684188
Title: Rural Options At Discharge Model of Active Planning
Acronym: ROADMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: Providence St. Patrick Hospital, Missoula Montana (Unknown)
Responsible Party: Principal Investigator, Tom Seekins, Professor of Psychology and Director, RTC:Rural, University of Montana
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 177-15
Record Dates: First submitted 2015-12-30; First posted 2016-02-17 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: All Causes Hospital Admissions

STUDY DESIGN:
Intervention Model Description: Patients were recruited from those admitted from one of four rural counties. In the initial phase, all patients enrolled from any county were assigned to a baseline condition. After enrollment stabilized, patients from one county were enrolled in the intervention while patients from the other three counties remained in baseline. Subsequently the intervention was introduced to the other counties sequentially while others remained in baseline. A return to baseline conditions followed a period after the intervention had been introduced in all counties.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard hospital discharge services (No Intervention): Patients received standard discharge planning; the baseline and return to baseline groups were combined to form a single standard discharge group
- Enhanced rural discharge and transition (Experimental): Enhanced rural discharge and transition involved conducting a functional needs assessment before discharge. Identified needs were shared with a Local Community Transition Coordinator (LCTC). Needs include such patient centered issues as housing, transportation, emotional support, support for completing daily chores, and assistance in securing local follow-up appointments. Once a patient returned home, the LCTC conduct a review of discharge orders to insure a patient can meet those recommendations. Then the LCTC worked with the patient to develop and implement a transition plan that linked the patient to local resources he or she can use to address needs. The LCTC also provided direct supports. This plan was implemented over the course of the first 30 days after discharge.
  Interventions: Behavioral: Enhanced rural discharge and transition

INTERVENTIONS:
Behavioral: Enhanced rural discharge and transition — While in the treating hospital, patients from small towns and rural communities are engaged in package of procedures designed to improve the transitions home, including a functional needs assessment that produces a plan that matches available rural community service providers to a patient's transitions needs and the provision of enhanced recovery supports to the patient.
  Arms: Enhanced rural discharge and transition

SUMMARY:
Residents of rural and frontier counties experience significant disparities in health care access and outcomes when compared to their urban counterparts. The organization of health care delivery contributes significantly to these disparities. For rural residents with multiple chronic conditions, transitioning along the continuum of care, between systems of treatment and support, and between dispersed locations present significant challenges. One critical challenge involves hospitalization for treatment because it requires travel to locations at a significant distance from home and disrupts personal and family routines. The transition back home is also problematic because discharge planning does not adequately account for limited access to care in rural areas. Indeed, discharge planning has been recently described as a "black hole;" fragmented and uncoordinated, and contributing to poor outcomes and patient dissatisfaction. The specific aim of this research is to ascertain rural patients' actual experience of the discharge planning process and to involve patients and rural providers in designing and testing a contextually appropriate rural options discharge model (ROADMAP) that improves patient outcomes and reduces re-hospitalizations.

DETAILED DESCRIPTION:
Residents of rural counties experience significant disparities in health care access and outcomes when compared to their urban counterparts. These disparities are structural; based in our market-based medical care delivery system. For rural residents with multiple chronic conditions, transitioning along the continuum of care, between systems of treatment and support, and between dispersed locations both expose and produce disparities. The transition home from hospitalization for treatment exposes the current urban bias. Indeed, discharge planning is fragmented and uncoordinated, and contributes to poor the disparities. The specific aims of this research is to ascertain rural patients' actual experience of discharge; then to involve patients and rural providers in using those data to design a contextually appropriate rural options at discharge model of active planning (ROADMAP) that improves patient outcomes and reduces disparities. Objectives include:

1. Ascertain actual patient experience in the rural discharge process.
2. Design the ROADMAP model to fit the emerging health services context.
3. Test the ROADMAP's efficacy in enhancing patient defined outcomes.
4. Design the components for rapid diffusion.

Researchers will work in four counties of the Missoula Hospital Referral Region with a total population of 53,116 living on 12,342 square miles (4.3 persons per square mile). Researchers will recruit patients seeking treatment from St. Patrick Hospital. Patients and patient advocates will serve on an Innovations Design Team (IDT) to create the ROADMAP. Researchers will first interview patients (n = 40) who have been discharged to one of the rural counties. Researchers will compare their experiences to guidelines. Next, they will conduct a Design Survey (n=600) to verify goals important to patients. The IDT will use these findings to develop design requirements for ROADMAP. Finally, we will use a quasi-experimental research design to compare the patient designed rural ROADMAP to standard practice. The primary outcome measures are measures that reflect the patient's values for health-related quality of life and functional status, as well as hospital re-admissions. An independent statistician will use Hierarchical Linear Modeling to examine the complex relationships. This approach accounts for patients nested in four counties and the correlated errors inherent in within subject analysis. Health care reform sets the occasion for rapid diffusion of ROADMAP. This can provide an incremental reduction in rural disparities. Incorporating patient and provider input increases the likelihood it will fit within the emerging reimbursement model. Researchers expect that ROADMAP will reduce re-hospitalizations by as much as 30%, and improve patient recovery and return to participation in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age
* Admitted to St. Patrick regional referral hospital for treatment
* Discharged home to one of four rural counties in Montana

Exclusion Criteria:

* Primary diagnosis involves psychiatric condition or substance abuse
* Inmates of state prison
* Admitted under ongoing criminal investigation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom W Seekins, Ph.D., Principal Investigator — University of Montana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants from among patients admitted to Saint Patrick Hospital, a regional referral hospital, from one of four counties. All four were non-metropolitan counties and three of the counties met the criteria of being a frontier county (population of less than 6 people per square mile).
Groups:
- Standard Hospital Discharge Planning Services: Patients receive standard discharge planning services.
- Enhanced Discharge Planning and Rural Transition Supports: The intervention consists of a package of procedures that enhances supports during the transitions from the hospital to recovery at home, including a structured needs assessment that produces a plan that matches available rural community service providers to a patient's transition needs and the provision of recovery supports to the patient.
  Enhanced Transitions Planning: While in the treating hospital, patients from small towns and rural communities are engaged in a process designed to improve the transitions home, including a functional needs assessment that produces a plan that matches available rural community service providers to a patient's transitions needs. Once home, a Local Community Transition Coordinator provides support to address needs.
Period: Overall Study
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Started | 77 | 50
Completed | 75 | 47
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Current Treatment: Patients receive that current discharge planning services and supports.
- Enhanced Transitions Planning: The intervention consists of a package of procedures that enhances supports during the transitions from the hospital to recovery at home, including a structured needs assessment that produces a plan that matches available rural community service providers to a patient's transitions needs and the provision of recovery supports to the patient.
  Enhanced Transitions Planning: While in the treating hospital, patients from small towns and rural communities are engaged in package of procedures designed to improve the transitions home, including a functional needs assessment that produces a plan that matches available rural community service providers to a patient's transitions needs and the provision of enhanced recovery supports to the patient.
- Total: Total of all reporting groups
Arm/Group | Current Treatment | Enhanced Transitions Planning | Total
Number analyzed (Participants) | 77 | 50 | 127
Age, Continuous [Mean (Full Range); unit: years] | 59.9 [30 to 74] | 63.2 [38 to 74] | 61.2 [30 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 21 | 55
  Male | 43 | 29 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 72 | 47 | 119
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 67 | 43 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants] — Participants recruited from among patients from four rural counties in St. Patrick Hospital's the catchment area, including Beaverhead, Lake, Powell, and Sanders Counties Montana.
  participants
    United States | 77 | 50 | 127
Patient Activation Measure (PAM10) [Mean (Full Range); unit: units on a scale] — Patients completed the 10-item Patient Activation Measure (PAM10) questionnaire measuring a patient's confidence in their knowledge, skills, and abilities to manage their health once they were discharged from a hospital. Patients indicated whether they strongly agreed, agreed, disagreed, or strongly disagreed with each statement. A patient could also indicate that a particular item was not applicable to their situation. Total scores ranged from 0.0 to 100.0. Higher scores indicated greater confidence in their capacity for self-management.
  units on a scale | 65.1 [39 to 100] | 73.8 [45 to 100] | 69.9 [39 to 100]
Length of Stay, Acuity, Co-morbidity, and Emergency Department Visits (LACE+) [Mean (Full Range); unit: units on a scale] — The LACE+ uses a proprietary algorithm to calculate the likelihood of a patient's hospital readmission based on information derived from the patient's electronic medical record. Generally, higher scores reflect higher risk. Scores range from 0 to 100. A score of 28 or less is categorized as low risk. A score of 29 to 58 is categorized as medium risk. A score of 59 or higher is categorized as high risk. Population: We analyzed LACE+ data for 112 patients as the electronic medical record did not establish this measure until after the study started.
  units on a scale
    number analyzed (Participants) | 62 | 50 | 112
    (all) | 42.2 [13 to 84] | 49.7 [22 to 80] | 46.3 [13 to 84]

OUTCOME MEASURES:

1. Primary Outcome: Hospital Re-admissions Analyzed by Poisson Regression
Description: Number of admissions to any hospital reported by the patients after discharge from a regional hospital to one of four rural counties.
Time Frame: 3, 7 ,14, 21, 30, 60, and 90 days after discharge
Population: Patients between 18 and 75 years old admitted to regional referral hospital for treatment, who enrolled in study and were discharged to one of four rural counties
Measure: Number; unit: Hospital Readmission
Groups:
- Enhanced Discharge & Rural Transition Support: The intervention consists of a package of procedures that enhances supports during the transitions from the hospital to recovery at home, including a structured needs assessment that produces a plan that matches available rural community service providers to a patient's transitions needs and the provision of recovery supports to the patient.
  Enhanced Discharge Planning & Rural Transition Support: While in the treating hospital, patients from small towns and rural communities are engaged in package of procedures designed to improve the transitions home, including a functional needs assessment that produces a plan that matches available rural community service providers to a patient's transitions needs and the provision of enhanced recovery supports to the patient.
Arm/Group | Standard Hospital Discharge Services | Enhanced Discharge & Rural Transition Support
Number analyzed (Participants) | 77 | 50
Hospital Readmission
  3 days after discharge | 17 | 4
  7 days after discharge | 21 | 5
  14 days after discharge | 23 | 7
  21 days after discharge | 25 | 7
  30 days after discharge | 25 | 9
  60 days after discharge | 28 | 10
  90 days after discharge | 26 | 12
Statistical Analysis 1: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 3 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 3; Test type: Superiority; p = 0.030, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 3, 112(68 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 2: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 7 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 7; Test type: Superiority; p = 0.025, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 7, 110 (66 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 3: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 14 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 14; Test type: Superiority; p = 0.037, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 14, 104 (61 baseline and 43 intervention) patients were used in this analysis
Statistical Analysis 4: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 21 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 21; Test type: Superiority; p = 0.011, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 21, 98 (57 baseline and 41 intervention) patients were used in this analysis
Statistical Analysis 5: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 30 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 30; Test type: Superiority; p = 0.050, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 30, 95 (56 baseline and 39 intervention) patients were used in this analysis
Statistical Analysis 6: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 60 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 60; Test type: Superiority; p = 0.055, Poisson regression; For day 60, 87 (53 baseline and 34 intervention) patients were used in this analysis
Statistical Analysis 7: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the cumulative number of hospital visits for day 90 (null hypothesis); H1: The cumulative number of hospital visits for the standard discharge group is greater than that for the enhanced discharge group for day 90; Test type: Superiority; p = 0.137, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 90, 83 (49 baseline and 34 intervention) patients were used in this analysis

2. Primary Outcome: Hospital Re-admissions Analyzed by Logistic Regression
Description: Proportion of patients who self-report at least one hospital readmission to any hospital after discharge from a regional hospital to one of four rural counties.
Time Frame: 3, 7 ,14, 21, 30, 60, and 90 days after discharge
Population: as for outcome 1
Measure: Number; unit: proportion of patients rehospitalized
Arm/Group | Standard Hospital Discharge Services | Enhanced Discharge & Rural Transition Support
Number analyzed (Participants) | 77 | 50
proportion of patients rehospitalized
  3 days after discharge: number analyzed (Participants) | 68 | 44
  3 days after discharge | 0.10 | 0.07
  7 days after discharge: number analyzed (Participants) | 66 | 44
  7 days after discharge | 0.12 | 0.07
  14 days after discharge: number analyzed (Participants) | 61 | 43
  14 days after discharge | 0.11 | 0.09
  21 days after discharge: number analyzed (Participants) | 57 | 41
  21 days after discharge | 0.16 | 0.10
  30 days after discharge: number analyzed (Participants) | 56 | 39
  30 days after discharge | 0.16 | 0.18
  60 days after discharge: number analyzed (Participants) | 53 | 34
  60 days after discharge | 0.19 | 0.18
  90 days after discharge: number analyzed (Participants) | 49 | 34
  90 days after discharge | 0.18 | 0.21
Statistical Analysis 1: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the proportion of patients with at least one ED visits by day 3 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 3; Test type: Superiority; p = 0.279, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 3, 112(68 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 2: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the proportion of patients with at least one ED visits by day 7 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 7; Test type: Superiority; p = 0.211, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 7, 110 (66 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 3: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the proportion of patients with at least one ED visits by day 14 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 14; Test type: Superiority; p = 0.424, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 14, 104 (61 baseline and 43 intervention) patients were used in this analysis
Statistical Analysis 4: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the proportion of patients with at least one ED visits by day 21 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 21; Test type: Superiority; p = 0.191, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 21, 98 (57 baseline and 41 intervention) patients were used in this analysis
Statistical Analysis 5: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the proportion of patients with at least one ED visits by day 30 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 30; Test type: Superiority; p = 0.478, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 30, 95 (56 baseline and 39 intervention) patients were used in this analysis
Statistical Analysis 6: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; H0: There is no difference in the proportion of patients with at least one ED visits by day 60 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 60; Test type: Superiority; p = 0.452, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 60, 87 (53 baseline and 34 intervention) patients were used in this analysis
Statistical Analysis 7: Comparison: Standard Hospital Discharge Services vs Enhanced Discharge & Rural Transition Support; Test type: Superiority — H0: There is no difference in the proportion of patients with at least one ED visits by day 90 (null hypothesis); H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 90; p = 0.381, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 90, 83 (49 baseline and 34 intervention) patients were used in this analysis

3. Primary Outcome: Emergency Department (ED) Visits Analyzed by Poisson Regression
Description: Number of self-reported visits to the emergency department of any hospital reported by patients after discharge from a regional hospital to one of four rural counties.
Time Frame: 3, 7, 14, 21,30, 60, and 90 days after discharge
Population: as for outcome 1
Measure: Number; unit: Emergency Department Visits
Groups:
- Standard Hospital Discharge Planning Services: Patients receive standard discharge planning services;the baseline and return to baseline groups were combined to form a single standard discharge group
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
Emergency Department Visits
  3 days after discharge: number analyzed (Participants) | 70 | 45
  3 days after discharge | 9 | 6
  7 days after discharge: number analyzed (Participants) | 68 | 45
  7 days after discharge | 18 | 11
  14 days after discharge: number analyzed (Participants) | 63 | 44
  14 days after discharge | 27 | 17
  21 days after discharge: number analyzed (Participants) | 59 | 42
  21 days after discharge | 38 | 19
  30 days after discharge: number analyzed (Participants) | 58 | 40
  30 days after discharge | 43 | 19
  60 days after discharge: number analyzed (Participants) | 55 | 35
  60 days after discharge | 47 | 19
  90 days after discharge: number analyzed (Participants) | 51 | 35
  90 days after discharge | 48 | 21
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.502, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 3, 115 (70 baseline and 45 intervention) patients were used in this analysis
Statistical Analysis 2: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of ED visits for day 7 (null hypothesis); H1: The cumulative number of ED visits for the standard discharge group is greater than that for the enhanced discharge group for day 7; Test type: Superiority; p = 0.286, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 7, 113 (68 baseline and 45 intervention) patients were used in this analysis
Statistical Analysis 3: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of ED visits for day 14 (null hypothesis); H1: The cumulative number of ED visits for the standard discharge group is greater than that for the enhanced discharge group for day 14; Test type: Superiority; p = 0.347, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 14, 107 (63 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 4: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of ED visits for day 21 (null hypothesis); H1: The cumulative number of ED visits for the standard discharge group is greater than that for the enhanced discharge group for day 21; Test type: Superiority; p = 0.250, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 21, 101 (59 baseline and 42 intervention) patients were used in this analysis
Statistical Analysis 5: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of ED visits for day 30 (null hypothesis); H1: The cumulative number of ED visits for the standard discharge group is greater than that for the enhanced discharge group for day 30; Test type: Superiority; p = 0.220, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 30, 98 (58 baseline and 40 intervention) patients were used in this analysis
Statistical Analysis 6: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of ED visits for day 60 (null hypothesis); H1: The cumulative number of ED visits for the standard discharge group is greater than that for the enhanced discharge group for day 60; Test type: Superiority; p = 0.116, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 60, 90 (55 baseline and 35 intervention) patients were used in this analysis
Statistical Analysis 7: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of ED visits for day 90 (null hypothesis); H1: The cumulative number of ED visits for the standard discharge group is greater than that for the enhanced discharge group for day 90; Test type: Superiority; p = 0.126, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 90, 86 (51 baseline and 35 intervention) patients were used in this analysis

4. Primary Outcome: Emergency Department (D) Visits Analyzed by Logistic Regression
Description: Proportion of patients who report at least one emergency department visit after discharge from a regional hospital to one of four rural counties.
Time Frame: 3, 7, 14, 21,30, 60, and 90 days after discharge
Population: as for outcome 1
Measure: Number; unit: participants with at least one ED visit
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
participants with at least one ED visit
  3 days after discharge: number analyzed (Participants) | 70 | 45
  3 days after discharge | 0.10 | 0.09
  7 days after discharge: number analyzed (Participants) | 68 | 45
  7 days after discharge | 0.15 | 0.11
  14 days after discharge: number analyzed (Participants) | 63 | 44
  14 days after discharge | 0.16 | 0.14
  21 days after discharge: number analyzed (Participants) | 59 | 42
  21 days after discharge | 0.22 | 0.19
  30 days after discharge: number analyzed (Participants) | 58 | 40
  30 days after discharge | 0.24 | 0.20
  60 days after discharge: number analyzed (Participants) | 55 | 35
  60 days after discharge | 0.29 | 0.23
  90 days after discharge: number analyzed (Participants) | 51 | 35
  90 days after discharge | .29 | 0.23
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 3; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 3; Test type: Superiority; p = 0.597, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 3, 115 (70 baseline and 45 intervention) patients were used in this analysis
Statistical Analysis 2: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 7; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 7; Test type: Superiority; p = 0.504, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 7, 113 (68 baseline and 45 intervention) patients were used in this analysis
Statistical Analysis 3: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 14; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 14; Test type: Superiority; p = 0.558, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 14, 107 (63 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 4: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 21; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 21; Test type: Superiority; p = 0.472, Regression, Logistic — Comments (covariates): P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 21, 101 (59 baseline and 42 intervention) patients were used in this analysis
Statistical Analysis 5: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 30; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 30; Test type: Superiority; p = 0.462, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 30, 98 (58 baseline and 40 intervention) patients were used in this analysis
Statistical Analysis 6: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 60; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 60; Test type: Superiority; p = 0.394, Regression, Logistic — P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 60, 90 (55 baseline and 35 intervention) patients were used in this analysis
Statistical Analysis 7: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the proportion of patients with at least one ED visits by day 90; H1: The proportion of patients with at least one ED visit for the standard discharge group is greater than that for the enhanced discharge group for day 90; Test type: Superiority; p = 0.368, Regression, Logistic — Comments (covariates): P-values comparing the counts for the 2 groups after adjusting for PAM10; For day 90, 86 (51 baseline and 35 intervention) patients were used in this analysis

5. Primary Outcome: Primary Care Provider (PCP) Visits Analyzed by Poisson Regression
Description: This reflects the number of visits to a patient's local primary care provider at 3, 7, 14, 21,30, 60, and 90 days after discharge.
Time Frame: 3, 7, 14, 21, 30, 60, and 90 days after discharge
Population: Patients between 18 and 75 years old admitted to a regional referral hospital for treatment, who enrolled in the study and were discharged to one of four rural counties.
Measure: Number; unit: Primary Care Provider Visits
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
Primary Care Provider Visits
  3 days after discharge: number analyzed (Participants) | 70 | 44
  3 days after discharge | 7 | 2
  7 days after discharge: number analyzed (Participants) | 67 | 44
  7 days after discharge | 27 | 19
  14 days after discharge: number analyzed (Participants) | 62 | 43
  14 days after discharge | 54 | 45
  21 days after discharge: number analyzed (Participants) | 58 | 40
  21 days after discharge | 71 | 50
  30 days after discharge: number analyzed (Participants) | 57 | 38
  30 days after discharge | 91 | 49
  60 days after discharge: number analyzed (Participants) | 54 | 33
  60 days after discharge | 135 | 59
  90 days after discharge: number analyzed (Participants) | 50 | 33
  90 days after discharge | 148 | 83
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; The following hypotheses were tested: H0: There is no difference in the cumulative number of PCP visits for day 3 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 3; Test type: Superiority; p = 0.946, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for sex, age, number in household, county, and LACE+ score; For day 3, 114 (70 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 2: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of PCP visits for day 7 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 7; Test type: Superiority; p = 0.613, Poisson regression; For day 7, 111 (67 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 3: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of PCP visits for day 14 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 14; Test type: Superiority; p = 0.541, Poisson regression — [p-value comment as in outcome 5, analysis 1]; For day 14, 105 (62 baseline and 43 intervention) patients were used in this analysis
Statistical Analysis 4: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of PCP visits for day 21 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 21; Test type: Superiority; p = 0.765, Poisson regression — P-values comparing the counts for the 2 groups after adjusting for sex, age, number in household, county, and LACE score; For day 21, 98 (58 baseline and 40 intervention) patients were used in this analysis
Statistical Analysis 5: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of PCP visits for day 30 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 30; Test type: Superiority; p = 0.919, Poisson regression — [p-value comment as in outcome 5, analysis 1]; For day 30, 95 (57 baseline and 38 intervention) patients were used in this analysis
Statistical Analysis 6: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of PCP visits for day 60 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 60; Test type: Superiority; p = 0.999, Poisson regression — [p-value comment as in outcome 5, analysis 4]; P-values comparing the counts for the 2 groups after adjusting for sex, age, number in household, county, and LACE score; For day 60, 87 (54 baseline and 33 intervention) patients were used in this analysis
Statistical Analysis 7: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; H0: There is no difference in the cumulative number of PCP visits for day 90 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 90; Test type: Superiority; p = 0.995, Poisson regression; For day 90, 83 (50 baseline and 33 intervention) patients were used in this analysis

6. Secondary Outcome: Short Form (SF12) Physical Health Score
Description: The SF12 is a twelve-item standardized questionnaire that measures overall, physical health, and mental health. Patients rate each item on an ordinal scale. Data are analyzed using a proprietary algorithm. Scores range from 0 to 100. Higher scores reflect a better health status. The analysis creates an overall health score and sub scores that reflect physical health and mental health. Both Physical and Mental Health Composite Scales combine the 12 items in such a way that they compare to a national norm of a mean score of 50.0 and a standard deviation of 10.0.
Time Frame: 3, 7, 14, 21, 30, 60, and 90 days after discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
units on a scale
  3 days after discharge | 35.1 (7.8) | 36.3 (7.9)
  7 days after discharge | 34.7 (6.6) | 35.1 (7.5)
  14 days after discharge | 35.7 (6.4) | 36.0 (6.7)
  21 days after discharge | 36.3 (6.1) | 36.4 (5.9)
  30 days after discharge | 37.3 (6.0) | 37.2 (7.1)
  60 days after discharge | 39.2 (5.8) | 39.0 (6.5)
  90 days after discharge | 40.3 (6.0) | 39.9 (6.1)
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; The following hypotheses were tested: Hoi: There is no difference in mean SF12 Physical Health scores between the standard and enhanced discharge groups (null hypothesis); H1i: The mean SF12 Physical Health scores differ between the standard and enhanced discharge groups; Test type: Equivalence — A repeated measures ANOVA model was used to model the SF12 Physical Health score as a function of treatment group. The likelihood ratio test was used to calculate the p-values for the treatment effect and covariates. No adjustments for multiple comparisons were made. Hypotheses were tested after adjusting for the effects of the repeated measures, patient age, and the number of people in a household. All hypotheses were 2-sided and p-values < 0.05 were considered statistically significant; p = 0.371, ANOVA — The P-value comparing the means for the 2 groups averaged across the 7 days is p = 0.371, after adjusting for covariates

7. Secondary Outcome: Short Form (SF12) Mental Health Score
Description: as for outcome 6
Time Frame: 3, 7, 14, 21, 30, 60, and 90 days after discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
units on a scale
  3 days after discharge | 47.8 (12.1) | 47.2 (11.2)
  7 days after discharge | 50.0 (12.5) | 49.3 (13.0)
  14 days after discharge | 51.8 (10.9) | 50.9 (10.5)
  21 days after discharge | 53.9 (10.6) | 54.5 (10.5)
  30 days after discharge | 53.8 (10.0) | 53.4 (11.0)
  60 days after discharge | 54.4 (8.7) | 53.6 (8.9)
  90 days after discharge | 54.8 (10.2) | 54.4 (9.2)
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; The following hypotheses were tested: Hoi: There is no difference in mean SF-12 Mental Health scores between the standard and enhanced discharge groups (null hypothesis); H1i: The mean SF-12 Mental Health scores differ between the standard and enhanced discharge groups; Test type: Equivalence — A repeated measures ANOVA model was used to model the SF-12 Mental Health score as a function of treatment group. The likelihood ratio test was used to calculate the p-values for the treatment effect and covariates. No adjustments for multiple comparisons were made. Hypotheses were tested after adjusting for the effects of the repeated measures, patient age, income, and county. All hypotheses were 2-sided and p-values < 0.05 were considered statistically significant; p = 0.232, ANOVA — The P-value comparing the means for the 2 groups averaged across the 7 days is p = 0.232, after adjusting for covariates

8. Secondary Outcome: Care Transition Measure (CTM3)
Description: The CTM3 is a three-item standardized questionnaire to measures patients' perspectives on coordination of hospital discharge care. Patients rate whether they strongly agree, agree, disagree, or strongly disagree with three items (hospital staff too my preferences into account, I had a good idea what I was responsible for once I left the hospital, and I clearly understood the purpose for taking each of my medications). They may also rate an items as not applicable to their situation. Ratings are converted to a scale that ranges from 0 to 100. Higher scores reflect better discharge care.
Time Frame: 3 days after discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Survey Response Scores
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 68 | 44
Survey Response Scores | 0.86 (0.18) | 0.80 (0.26)
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; The following hypotheses were tested: H0: There is no difference in the mean CTM3 score between the standard and enhanced discharge groups (null hypothesis); H1: Patients in the enhanced discharge group will have a higher mean CTM3 rating than patients in the standard discharge group; Test type: Superiority; p = 0.806, ANCOVA; An analysis of covariance was used to model the CTM3 discharge planning score as a function of treatment group. An ANOVA F-test was used to calculate the p-values for the treatment effect and covariates. No adjustments for multiple comparisons were made. Hypotheses were tested after adjusting for the effects of patient age and income. The hypothesis test for the group comparison was 1-sided, hypotheses to assess significance of covariates were 2-sided, and p-values < 0.05 were considered statistically significant. The covariates Sex, County, Number in Household, LACE+ score, and PAM10 score did not differ in their mean CTM3 scores so were not retained in the model

9. Secondary Outcome: Rural Transition Measure (RTM14)
Description: The RTM14 is a fourteen-item questionnaire to measures patients' perspectives on the delivery of transition services and supports after discharge from a regional hospital to a small town or rural community. Patients respond by indicating whether they strongly disagree, disagree, agree, or strongly agree with each of the 14 items. Patients may also indicate whether an item is not applicable to their situation. Ratings are converted to a scale that ranges from 0 to 100. Higher scores reflect better transition service performance.
Time Frame: 7, 14, 21, 30, 60, and 90 days after discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Survey Response Scores
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
Survey Response Scores
  7 days after discharge | 0.854 (0.173) | 0.884 (0.149)
  14 days after discharge | 0.897 (0.131) | 0.873 (0.161)
  21 days after discharge | 0.922 (0.118) | 0.876 (0.158)
  30 days after discharge | 0.902 (0.133) | 0.895 (0.147)
  60 days after discharge | 0.901 (0.120) | 0.924 (0.092)
  90 days after discharge | 0.901 (0.163) | 0.911 (0.107)
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; The following hypotheses were tested: H0: There is no difference in the mean RTM14 score between the standard and enhanced discharge groups (null hypothesis); H1: Patients in the enhanced discharge group will have a higher mean RTM14 rating than patients in the standard discharge group; Test type: Superiority; p = 0.742, ANOVA; A repeated measures ANOVA model (over the 6 time measurement periods) was used to model the RTM14 score as a function of treatment group. The likelihood ratio test was used to calculate the p-values for the treatment effect and covariates. No adjustments for multiple comparisons were made. Hypotheses were tested after adjusting for the effects of the repeated measures, patient age, income, and whether or not a patient had visited a hospital or ED prior to that day. The hypothesis test for the group comparison was 1-sided, hypotheses to assess significance of covariates were 2-sided, and p-values < 0.05 were considered statistically significant. The covariates Sex, Number in household, LACE+ score, and PAM10 score were not significant in explaining SF-12 scores so were not retained in the model

10. Primary Outcome: Primary Care Provider (PCP) Visits Analyzed by Logistic Regression
Description: This reflects the proportion of patients who reported at least one visit to a their local primary care provider at 3, 7, 14, 21,30, 60, and 90 days after discharge.
Time Frame: 3, 7, 14, 21, 30, 60, and 90 days after discharge
Population: as for outcome 5
Measure: Number; unit: Proportion with Primary Care Visits
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
Number analyzed (Participants) | 77 | 50
Proportion with Primary Care Visits
  3 days after discharge: number analyzed (Participants) | 70 | 44
  3 days after discharge | 0.07 | 0.05
  7 days after discharge: number analyzed (Participants) | 67 | 44
  7 days after discharge | 0.31 | 0.32
  14 days after discharge: number analyzed (Participants) | 62 | 43
  14 days after discharge | 0.47 | 0.51
  21 days after discharge: number analyzed (Participants) | 58 | 40
  21 days after discharge | 0.60 | 0.53
  30 days after discharge: number analyzed (Participants) | 57 | 38
  30 days after discharge | 0.63 | 0.55
  60 days after discharge: number analyzed (Participants) | 54 | 33
  60 days after discharge | 0.74 | 0.64
  90 days after discharge: number analyzed (Participants) | 50 | 33
  90 days after discharge | 0.80 | 0.70
Statistical Analysis 1: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; : H0: There is no difference in the cumulative number of PCP visits for day 3 (null hypothesis); H1: The cumulative number of PCP visits for the standard discharge group is less than that for the enhanced discharge group for day 3; Test type: Superiority; p = 0.717, Regression, Logistic — This Hypothesis was tested with no adjustments for covariates since none were significant; For day 3, 114 (70 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 2: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.479, Regression, Logistic — This Hypothesis was tested with no adjustments for covariates since none were significant; For day 7, 111 (67 baseline and 44 intervention) patients were used in this analysis
Statistical Analysis 3: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.329, Regression, Logistic; For day 14, 105 (62 baseline and 43 intervention) patients were used in this analysis
Statistical Analysis 4: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.780, Regression, Logistic; This Hypothesis was tested with no adjustments for covariates since none were significant
Statistical Analysis 5: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.779, Regression, Logistic — This Hypothesis was tested with no adjustments for covariates since none were significant; For day 30, 95 (57 baseline and 38 intervention) patients were used in this analysis
Statistical Analysis 6: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.848, Regression, Logistic — This Hypothesis was tested with no adjustments for covariates since none were significant; For day 60, 87 (54 baseline and 33 intervention) patients were used in this analysis
Statistical Analysis 7: Comparison: Standard Hospital Discharge Planning Services vs Enhanced Discharge Planning and Rural Transition Supports; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.857, Regression, Logistic — This Hypothesis was tested with no adjustments for covariates since none were significant; For day 90, 83 (50 baseline and 33 intervention) patients were used in this analysis

ADVERSE EVENTS:
Time Frame: Up to 90 days post discharge
Arm/Group | Standard Hospital Discharge Planning Services | Enhanced Discharge Planning and Rural Transition Supports
All-Cause Mortality (participants affected / at risk) | 2/77 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/50
Other Adverse Events (participants affected / at risk) | 0/77 | 0/50

LIMITATIONS AND CAVEATS:
The overall sample was small due to the rural focus of the program. The sample size for emergency department visits and hospitalizations was low, making it difficult to detect differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT02684188/Prot_SAP_000.pdf